CLINICAL TRIAL: NCT03550560
Title: Drainage of Refractory Malignant Ascites by Endoscopic Ultrasound-guided (EUS-Guided) Implantation of Plastic Prostheses
Brief Title: EUS-Guided Drainage of Refractory Malignant Ascites
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitario Virgen Macarena (Other)
Collaborators: Delos Clinical (Other)
Responsible Party: Sponsor
Other Study IDs: JBO-ECO-2017-01
Record Dates: First submitted 2018-03-15; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Malignant Ascites
Keywords: Endoscopic Ultrasound-Guided; EUS-Guided; Transgastric plastic prostheses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- EUS-Guided drainage: Cancer patients in terminal phase with refractory malignant ascites
  Interventions: Procedure: EUS-Guided drainage

INTERVENTIONS:
Procedure: EUS-Guided drainage — Drainage of refractory malignant ascites by endoscopic ultrasound-guided (EUS-Guided) implantation of plastic prostheses.

SUMMARY:
This study evaluates the efficacy and safety of drainage of refractory malignant ascites by endoscopic ultrasound-guided (EUS-Guided) implantation of plastic prostheses. Patients with cancer older than 18 years with a life expectancy of less than 6 months who undergo EUS-Guided will be included in the study.

DETAILED DESCRIPTION:
Malignant ascites is described as the presence of fluid in the abdominal cavity due to the presence of tumors. Its appearance is a predictor of worse prognosis in the evolution of malignant neoplasm and reduces the quality of life of patients.

The use of prostheses with drainage to the gastric cavity has shown good clinical results as the reduction of paracentesis evacuation needs. This achieves the reduction of hospital admissions and the improvement of the quality of life of the patient.

In order to verify the usefulness of this drainage technique, a prospective observational study has been designed. Patients with cancer over 18 years of age will be included, with a life expectancy of less than 6 months and who have undergone drainage of refractory malignant ascites through the implantation of plastic prostheses.

Participants receive the intervention in the same manner and intensity if they are not enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients in terminal phase with refractory malignant ascites older 18 years of age

Exclusion Criteria:

* Patients under 18 years of age
* Patients with a life expectancy greater than 6 months
* Patients who are receiving cancer treatment for curative purposes or who suffer from a psychiatric disorder that prevents them from understanding and accepting the procedure
* Patients who do not accept to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients in terminal phase with refractory malignant ascites
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of new evacuation paracentesis after the procedure. | At 1 week.
  Paracentesis is an invasive technique that, by means of an abdominal percutaneous puncture, allows us to evacuate fluid from the peritoneal cavity. However, it only provides temporary improvement because the rapid recurrence of fluid usually occurs in about 72 hours.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0. | At 1 week.
  CTCAE is widely accepted throughout the oncology community as the standard classification and severity grading scale for adverse events in cancer therapy clinical trials and other oncology settings.
Change in quality of life by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 15-palliative care (EORTC QLQ-C15-PAL) | From baseline at 1 week.
  EORTC QLQ-C15-PAL is a questionnaire developed to assess the quality of life of palliative cancer care patients. It comprises 15 questions including two functional scales (physical function and emotional function), two multi-item symptom scales (fatigue and pain), and five single-item symptom scales (nausea and vomiting, dyspnea, insomnia, appetite loss, and constipation). Response options to these 14 items use a four-point Likert scale: 1 (not at all), 2 (a little), 3 (quite a bit), and 4 (very much). An additional item, global health/quality-of-life scale, uses a seven point numerical scale from 1 (very poor) to 7 (excellent). Higher scores for the functional scale and global health/quality-of-life scale indicate better quality of life. However, higher symptom scales indicate lower quality of life.
Change in Dyspnea by The modified Medical Research Council (mMRC) Scale. | From baseline at 1 week.
  The mMRC scale is used to establish the severity of dyspnea attributable to the respiratory disease.
  The mMRC is a self-administered questionnaire where the patient must choose one among five statements based on the perception of the patient in daily activities:
  0. Not troubled by breathlessness except on strenuous exercise.
  1. Short of breath when hurrying or walking up a slight hill.
  2. Walks slower than peers on level ground due to dyspnea, or must to stop for breath when walking at own pace.
  3. Stops for breath after walking about 100m or after a few minutes on level ground.
  4. Too breathless to leave the house, or breathless when dressing or undressing.
  According to the patient's response, dyspnea is classified as: 0. None, 1. Mild, 2. Moderate, 3. Severe and 4. Very severe.
Change in abdominal pain by The Visual Analogue Scale (VAS). | From baseline at 1 week.
  VAS is a measurement instrument that permite to measure pain. The VAS used is a straight horizontal line of 100 mm. The ends are defined as the extreme limits of the parameter to be measured orientated from the left (worst) to the right (best). Using a ruler, the score is determined by measuring the distance (mm) between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Change in abdominal circumference. | From baseline at 1 week.
  Circumference in centimeters.
Change in weight. | Form baseline at 1 week.
  Weight in kilograms.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Romero Castro, Dr., Principal Investigator — Hospital Universitario Virgen Macarena

IPD SHARING:
Plan to Share IPD: Undecided